CLINICAL TRIAL: NCT07069075
Title: The Relationship Between MMP-2 and TIMP-2 Gene Polymorphisms and Skin Barrier Function, Inflammatory Cytokine Levels in Acne Patients
Brief Title: Gene Polymorphisms, Skin Barrier, and Inflammation in Acne
Status: Completed | Type: Observational
Sponsor: Hong Zhang (Other)
Responsible Party: Sponsor-Investigator, Hong Zhang, Principal investigator, Shijiazhuang TCM Hospital
Organization: Shijiazhuang TCM Hospital (Other)
Other Study IDs: 2020SJZTCMLL-KY0045
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Acne Vulgaris
Keywords: Acne; MMP-2; TIMP-2; Gene Polymorphism
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples were collected from all participants. Genomic DNA was extracted from whole blood for genotyping of MMP-2 rs243865 and TIMP-2 rs8179090. Serum was separated for measuring inflammatory cytokine levels (IL-1β, TNF-α) via ELISA.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acne Patients: Individuals aged 18 years or older who were diagnosed with acne vulgaris by a dermatologist. Participants provided blood samples for genotyping and cytokine analysis, and underwent non-invasive skin function tests.
  Interventions: Genetic: MMP-2 Gene Polymorphism (rs243865) Analysis; Genetic: TIMP-2 Gene Polymorphism (rs8179090) Analysis
- Healthy Controls: Healthy volunteers aged 18 years or older without any systemic or skin diseases, recruited during the same period. Participants provided blood samples for genotyping.
  Interventions: Genetic: MMP-2 Gene Polymorphism (rs243865) Analysis; Genetic: TIMP-2 Gene Polymorphism (rs8179090) Analysis

INTERVENTIONS:
Genetic: MMP-2 Gene Polymorphism (rs243865) Analysis — Participants were genotyped for the MMP-2 rs243865 polymorphism. Genomic DNA was extracted from peripheral blood, and the specific genotype (CC, CT, or TT) was determined using Polymerase Chain Reaction-Restriction Fragment Length Polymorphism (PCR-RFLP) analysis. This allowed for the stratification of participants based on their genetic variation at this locus for subsequent association analysis.
Genetic: TIMP-2 Gene Polymorphism (rs8179090) Analysis — Participants were genotyped for the TIMP-2 rs8179090 polymorphism. Genomic DNA was extracted from peripheral blood, and the specific genotype (CC, GC, or GG) was determined using Polymerase Chain Reaction-Restriction Fragment Length Polymorphism (PCR-RFLP) analysis. This allowed for the stratification of participants based on their genetic variation at this locus for subsequent association analysis.

SUMMARY:
This study investigated the relationship between Matrix Metalloproteinase-2 (MMP-2) and Tissue Inhibitor of Metalloproteinase-2 (TIMP-2) gene polymorphisms and acne pathogenesis. The study aimed to determine whether specific genotypes (MMP-2-CC and TIMP-2-CC) are associated with impaired skin barrier function (measured by transepidermal water loss and skin hydration) and elevated levels of inflammatory cytokines (IL-1β, TNF-α) in acne patients compared to healthy controls.

DETAILED DESCRIPTION:
Acne vulgaris is a common dermatological condition with a complex pathogenesis involving skin barrier dysfunction and inflammation. Matrix metalloproteinases (MMPs) and their tissue inhibitors (TIMPs) are crucial in extracellular matrix remodeling and have been implicated in acne. This case-control study was designed to explore the association of specific polymorphisms in the MMP-2 (rs243865) and TIMP-2 (rs8179090) genes with clinical and biological markers in acne. A total of 200 acne patients and 100 healthy controls were enrolled. Genomic DNA was extracted from peripheral blood samples, and genotyping was performed using PCR-RFLP. Skin barrier function was assessed by measuring Transepidermal Water Loss (TEWL) and skin hydration. Serum levels of the inflammatory cytokines Interleukin-1β (IL-1β) and Tumor Necrosis Factor-α (TNF-α) were quantified using ELISA. The study evaluates whether the CC genotypes of MMP-2 and TIMP-2 are risk factors for acne susceptibility and are correlated with more severe disease phenotypes, characterized by poorer skin barrier integrity and a heightened inflammatory state.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older, regardless of gender.
* Diagnosed with acne by a dermatologist (for patient group).
* No systemic or skin diseases (for control group).
* Able to provide informed consent and willing to undergo genotype testing and related skin function tests.

Exclusion Criteria:

* Acne induced by medications.
* Polycystic ovary syndrome or other forms of hormone-related acne.
* Any local, systemic, or surgical acne/acne scar treatments within the last four weeks.
* Presence of genetic connective tissue diseases.
* Associated with pyoderma or other systemic comorbidities.
* Refusal to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with acne vulgaris and healthy volunteers recruited from the dermatology department of Shijiazhuang TCM Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Genotype Frequencies of MMP-2 and TIMP-2 | Data for each participant were collected at a single visit during the study period from March 2018 to September 2021.
  Comparison of the genotype distribution (CC vs. CT/TT for MMP-2; CC vs. GC/GG for TIMP-2) between acne patients and healthy controls to assess association with acne susceptibility. [Time Frame: Data collected at a single study visit] Skin Barrier Function Assessment: Measurement of Transepidermal Water Loss (TEWL) and skin hydration levels in acne patients, compared across different MMP-2 and TIMP-2 genotypes.
Skin Barrier Function Assessment | Data for each participant were collected at a single visit during the study period from March 2018 to September 2021.
  Measurement of Transepidermal Water Loss (TEWL) and skin hydration levels in acne patients, compared across different MMP-2 and TIMP-2 genotypes.
Serum Interleukin-1β (IL-1β) Level | Data for each participant were collected at a single visit during the study period from March 2018 to September 2021.
  Measurement of serum levels of IL-1β in acne patients, compared across different MMP-2 and TIMP-2 genotypes.
Serum Tumor Necrosis Factor-α (TNF-α) Level | Data for each participant were collected at a single visit during the study period from March 2018 to September 2021.
  Measurement of serum levels of TNF-α in acne patients, compared across different MMP-2 and TIMP-2 genotypes.

SECONDARY OUTCOMES:
Correlation Analysis | Analysis was performed after the completion of data collection in September 2021.
  Pearson correlation and logistic regression analyses to evaluate the association between the MMP-2/TIMP-2 genotypes, impaired skin barrier function, and elevated inflammatory cytokine levels in acne patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Shijiazhuang TCM Hospital, Shijiazhuang, Hebei, China